CLINICAL TRIAL: NCT01306617
Title: An Open-Label Pilot Study to Evaluate the Antiviral Activity, Safety and Pharmacokinetics of ABT-450 With Ritonavir (ABT-450/r) Dosed in Combination With ABT-333 and Ribavirin (RBV) in Treatment-Naive and Non-responder Subjects With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of ABT-450 With Ritonavir (ABT-450/r) When Given Together With ABT-333 and Ribavirin (RBV) in Treatment-Naïve and Non-responder Subjects With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M12-746
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Results first posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Hepatitis C Infection; Hepatitis C; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — paritaprevir; dasabuvir; Ribavirin; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ABT-450/r (250/100 mg) and ABT-333 plus RBV in treatment-naïve (Experimental): ABT-450/r (250/100 mg) once daily (QD) and ABT-333 (400 mg) twice daily (BID) plus weight-based ribavirin (RBV) divided BID for 12 weeks in treatment-naïve participants.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ribavirin; Drug: ritonavir
- ABT-450/r (150/100 mg) and ABT-333 plus RBV in treatment-naïve (Experimental): ABT-450/r (150/100 mg) once daily (QD) and ABT-333 (400 mg) twice daily (BID) plus weight-based ribavirin (RBV) divided BID for 12 weeks in treatment-naïve participants.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ribavirin; Drug: ritonavir
- ABT-450/r (150/100 mg) and ABT-333 plus RBV in non-responders (Experimental): ABT-450/r (150/100 mg) once daily (QD) and ABT-333 (400 mg) twice daily (BID) plus weight-based ribavirin (RBV) divided BID in previous non-responders to pegylated interferon (pegIFN) and RBV.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ribavirin; Drug: ritonavir

INTERVENTIONS:
Drug: ABT-450 — tablets
Drug: ABT-333 — tablets
  Other Names: dasabuvir
Drug: ribavirin — tablets
Drug: ritonavir — capsules
  Other Names: Norvir

SUMMARY:
The purpose of this study is to evaluate the antiviral activity, safety, and pharmacokinetics of ABT-450 with ritonavir (ABT-450/r) dosed in combination with ABT-333 (also known as dasabuvir) and ribavirin (RBV) in treatment-naïve and non responder participants with genotype 1 chronic hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
This was a phase 2a multicenter, open-label, sequential, 3-arm, combination treatment study of a regimen of ABT-450/r/ABT-333, and ribavirin (RBV) in hepatitis C virus (HCV) genotype 1-infected treatment-naïve participants and previous non-responders to pegylated interferon (pegIFN)/RBV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C virus (HCV)
* Treatment naive, null or partial responders to previous treatment with peginterferon and ribavirin
* Males and females 18-65 years old
* Body mass index 18 to < 35 kg/m^2
* Females must be postmenopausal for at least 2 years or surgically sterile

Exclusion Criteria:

* Cirrhosis or extensive bridging fibrosis
* History of cardiac disease
* Positive screen for certain drugs or alcohol
* Abnormal laboratory results
* Significant sensitivity to any drug
* Positive hepatitis B surface antigen or anti-human immunodeficiency virus antibody
* Use of strong cytochrome P450 3A (CYP3A), cytochrome P450 2C8 (CYP2C8), and organic anion transporting polypeptide 1B1 (OATP1B1) enzyme inducers or inhibitors within 1 month of dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, MD, Study Director — AbbVie
Locations (11):
- United States (11):
  - Site Reference ID/Investigator# 48263, Los Angeles, California
  - Site Reference ID/Investigator# 48264, Aurora, Colorado
  - Site Reference ID/Investigator# 51282, Gainesville, Florida
  - Site Reference ID/Investigator# 50425, Springfield, Massachusetts
  - Site Reference ID/Investigator# 50423, Kansas City, Missouri
  - Site Reference ID/Investigator# 48268, New York, New York
  - Site Reference ID/Investigator# 50428, Statesville, North Carolina
  - Site Reference ID/Investigator# 48266, San Antonio, Texas
  - Site Reference ID/Investigator# 50427, Newport News, Virginia
  - Site Reference ID/Investigator# 48265, Seattle, Washington
  - Site Reference ID/Investigator# 50424, Madison, Wisconsin

REFERENCES:
- [Derived] Poordad F, Lawitz E, Kowdley KV, Cohen DE, Podsadecki T, Siggelkow S, Heckaman M, Larsen L, Menon R, Koev G, Tripathi R, Pilot-Matias T, Bernstein B. Exploratory study of oral combination antiviral therapy for hepatitis C. N Engl J Med. 2013 Jan 3;368(1):45-53. doi: 10.1056/NEJMoa1208809. PMID 23281975
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Started | 19 | 14 | 17
Completed | 18 (The number of participants who completed study drug) | 13 (The number of participants who completed study drug) | 12 (The number of participants who completed study drug)
Not Completed | 1 | 1 | 5
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Virologic Failure | 0 | 0 | 5
Not completed — Non-compliance | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analyses included all participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders | Total
Number analyzed (Participants) | 19 | 14 | 17 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (9.78) | 50.9 (10.45) | 52.3 (9.03) | 52.4 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 6 | 15
  Male | 10 | 14 | 11 | 35
Hepatitis C Virus (HCV) Genotype/ Subtype [Number; unit: participants]
  1A | 17 | 11 | 16 | 44
  1B | 2 | 3 | 1 | 6
Interleukin 28B (IL28B) Genotype [Number; unit: participants]
  CC | 10 | 5 | 0 | 15
  CT | 7 | 7 | 12 | 26
  TT | 2 | 2 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Suppressed Below the Lower Limit of Detection (LLOD) From Week 4 Through Week 12
Description: Analysis of the percentage of participants with hepatitis C virus ribonucleic acid less than the lower limit of detection (< 15 IU/mL).
Time Frame: Week 4 through Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT). Participants with missing data were imputed as failures.
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 19 | 14 | 17
percentage of participants | 89.5 | 78.6 | 58.8
Statistical Analysis 1: Comparison: ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve; For the percentage of subjects with HCV RNA suppressed below the LLOD from Week 4 through Week 12, if it was assumed that 60% of subjects would be successfully suppressed from Week 4 through Week 12, then 20 subjects in arm 1 would give a 95% 2-sided confidence interval (CI) of (38.5%, 81.5%), 10 subjects in arm 2 would give a 95% CI of (29.6%, 90.4%), and 15 subjects in arm 3 would give a 95% CI of (35.2%, 84.8%) for the percentage of subjects suppressed using the binomial exact method; Test type: Superiority or Other; p = 0.547, Regression, Logistic; Arm, baseline log10 HCV RNA level (<=800,000, >800,000), IL-28B genotype (CC, non-CC), and HCV subgenotype (1a, 1b) were used as strata
Statistical Analysis 2: Comparison: ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders; Test type: Superiority or Other; p = 0.207, Regression, Logistic; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants With HCV RNA < 1000 International Units Per Milliliter (IU/mL)
Description: Analysis of participants with HCV RNA levels below 1000 IU/mL at Week 2.
Time Frame: Week 2
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 19 | 14 | 17
percentage of participants | 100 | 92.9 | 100
Statistical Analysis 1: Comparison: ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve; Test type: Superiority or Other; p = 0.061, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With HCV RNA Below the Lower Limit of Quantitation (LLOQ; <25 IU/mL) at Week 4
Description: Analysis of percentage of participants with hepatitis C virus ribonucleic acid less than the lower limit of quantitation (< 25 IU/mL).
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 19 | 14 | 17
percentage of participants | 100 | 92.9 | 88.2
Statistical Analysis 1: Comparison: ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve; Test type: Superiority or Other; p = 0.061, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders; Test type: Superiority or Other; p = 0.375, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks (SVR12) Post-treatment
Description: Sustained virologic response 12 (SVR12) is defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (LLOQ; < 25 IU/mL) 12 weeks after the last dose of study drug.
Time Frame: Post-treatment Day 1 to Post-treatment Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 19 | 14 | 17
percentage of participants | 94.7 | 92.9 | 47.1
Statistical Analysis 1: Comparison: ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve; Test type: Superiority or Other; p = 0.312, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders; Test type: Superiority or Other; p = 0.012, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks (SVR24) Post-Treatment
Description: Sustained virologic response 24 (SVR24) is defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) less than the lower limit of quantification (LLOQ; < 25 IU/mL) 24 weeks after the last dose of study drug.
Time Frame: Post-treatment Day 1 to Post-treatment Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 19 | 14 | 17
percentage of participants | 94.7 | 85.7 | 47.1
Statistical Analysis 1: Comparison: ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve; Test type: Superiority or Other; p = 0.312, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders; Test type: Superiority or Other; p = 0.012, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Time to Failure to Suppress or Rebound During Treatment
Description: Time to failure to achieve a 2 log10 IU/mL HCV RNA decrease at Week 1, failure to achieve HCV RNA < Lower Limit of Detection (LLOD) at Week 6, or a confirmed increase of at least 0.5 log10 IU/mL above nadir (local minimum value) or confirmed HCV RNA > lower limit of quantitation (LLOQ) for participants who previously achieved HCV RNA < LLOQ.
Time Frame: Day 1 through Week 12
Population: Efficacy analyses included all participants who received at least 1 dose of study drug (ITT).
Measure: Mean (Standard Error); unit: days
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 19 | 14 | 17
days | 43.0 (NA) — Cannot be estimated as only one participant experienced virologic failure during treatment. | NA (NA) — Mean and standard error cannot be estimated as no participants experienced virologic failure during treatment in this arm. | 62.6 (5.44)
Statistical Analysis 1: Comparison: ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve; Test type: Superiority or Other; p = 0.395, Log Rank
Statistical Analysis 2: Comparison: ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders; Test type: Superiority or Other; p = 0.010, Log Rank

7. Secondary Outcome: Time to Virologic Relapse Post-treatment
Description: Time to the first of 2 consecutive measurements of confirmed HCV RNA ≥ lower limit of quantitation (LLOQ) at any point in the post-treatment period among participants with HCV RNA < LLOQ at the end of treatment.
Time Frame: Post-treatment Day 1 to post-treatment week 48
Population: All randomized participants who received at least 1 dose of study drug with HCV RNA < LLOQ at the final treatment visit who completed treatment.
Measure: Mean (Standard Error); unit: days
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 18 | 13 | 11
days | NA (NA) — Mean and standard error cannot be estimated as no participants experience relapse in this arm. | NA (NA) — Mean and standard error cannot be estimated as no participants experience relapse in this arm. | 15.8 (0.21)
Statistical Analysis 1: Comparison: ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve vs ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders; Test type: Superiority or Other; p = 0.048, Log Rank

8. Secondary Outcome: Resistance-Associated Variants and Phenotypic Resistance
Description: Baseline samples were analyzed for resistance-associated amino acid variants using population sequencing. Phenotypic resistance to ABT-450 or ABT-333 at baseline was assessed by calculating the fold difference in the half maximal effective concentration (EC50) compared with the EC50 for the appropriate reference replicon (1a-H77 or 1b-Con1). Participants not achieving SVR12 were analyzed for resistance-associated variants at the time of failure using population sequencing and were compared with the baseline and appropriate reference sequences to assess amino acid changes. Phenotypic resistance to ABT-450 or ABT-333 at the time of failure was assessed by calculating the fold difference in the EC50 compared with the EC50 for the corresponding baseline sample. The number of participants with variants at resistance-associated amino acid positions and phenotypic resistance at baseline and at the time of failure are presented.
Time Frame: Day 1 to post-treatment week 48
Population: Resistance analyses included all participants who receive at least one dose of study drug (intent-to-treat [ITT] population).
Measure: Number; unit: participants
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 19 | 14 | 17
participants
  Baseline Variants in NS3; n=49 | 0 | 0 | 1
  Baseline Resistance to ABT-450 >10-fold; n=40 | 0 | 0 | 1
  Baseline Variants in NS5B; n=49 | 2 | 2 | 0
  Baseline Resistance to ABT-333 >10-fold; n=49 | 0 | 1 | 0
  Post-treatment resistant variants in NS3; n=11 | 0 | 0 | 8
  Post-treatment resistance to ABT-450 >10-fold; n=9 | 0 | 0 | 6
  Post-treatment resistant variants in NS5B; n=11 | 0 | 0 | 8
  Post-treatment resistance to ABT-333 >10-fold;n=11 | 0 | 0 | 8

9. Secondary Outcome: Pharmacokinetics (C Trough) of ABT 450 in HCV Infected Participants
Description: Trough concentration (C trough) is the concentration 24 hours after once daily (QD) dose and 12 hours after twice daily (BID) dose.
Time Frame: Day 1 to Week 12
Population: Pharmacokinetic analyses included all participants who received at least 1 dose of the study drug (ITT) and for whom concentration data was available to characterize C trough.
Measure: Geometric Mean (Full Range); unit: nanograms (ng) per milliliter (mL)
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 14 | 11 | 9
nanograms (ng) per milliliter (mL) | 53.21 [4.64 to 1978.89] | 16.81 [2.70 to 191.23] | 16.15 [2.33 to 174.60]

10. Secondary Outcome: Pharmacokinetics (C Trough) of ABT-333 in HCV Infected Participants
Description: as for outcome 9
Time Frame: Day 1 to Week 12
Population: as for outcome 9
Measure: Geometric Mean (Full Range); unit: nanograms (ng) per milliliter (mL)
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 14 | 11 | 10
nanograms (ng) per milliliter (mL) | 148.44 [50.04 to 816.89] | 162.57 [76.92 to 579.67] | 166.15 [89.80 to 527.00]

11. Secondary Outcome: Pharmacokinetics (C Trough) of Ritonavir in HCV Infected Participants
Description: as for outcome 9
Time Frame: Day 1 to Week 12
Population: as for outcome 9
Measure: Geometric Mean (Full Range); unit: nanograms (ng) per milliliter (mL)
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 14 | 11 | 9
nanograms (ng) per milliliter (mL) | 43.92 [9.45 to 384.88] | 42.35 [12.07 to 1099.40] | 44.21 [23.73 to 73.76]

12. Secondary Outcome: Pharmacokinetics (C Trough) of Ribavirin in HCV Infected Participants
Description: as for outcome 9
Time Frame: Day 1 to Week 12
Population: as for outcome 9
Measure: Geometric Mean (Full Range); unit: nanograms (ng) per milliliter (mL)
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naïve | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Number analyzed (Participants) | 14 | 11 | 10
nanograms (ng) per milliliter (mL) | 2480 [1100 to 4800] | 2280 [1580 to 3760] | 2000 [1210 to 3880]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of study drug administration to 30 days after last dose of study drug (16 weeks).
Description: Serious Adverse Events (SAEs) were also collected from the time that informed consent was obtained through the end of the study (approximately 64 weeks).
Groups:
- ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naive: ABT-450/r (250/100 mg) once daily (QD) and ABT-333 (400 mg) twice daily (BID) plus weight-based ribavirin (RBV) divided BID for 12 weeks in treatment-naïve participants.
- ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naive: ABT-450/r (150/100 mg) once daily (QD) and ABT-333 (400 mg) twice daily (BID) plus weight-based ribavirin (RBV) divided BID for 12 weeks in treatment-naïve participants.
Arm/Group | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naive | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naive | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/14 | 0/17
Other Adverse Events (participants affected / at risk) | 17/19 | 13/14 | 13/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r (250/100 mg) and ABT-333 Plus RBV in Treatment-naive (N=19) | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Treatment-naive (N=14) | ABT-450/r (150/100 mg) and ABT-333 Plus RBV in Non-responders (N=17)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 1 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 1
EYE HAEMORRHAGE (Eye disorders) | 0 | 0 | 1
LACRIMATION INCREASED (Eye disorders) | 1 | 0 | 0
PHOTOPHOBIA (Eye disorders) | 0 | 1 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0
CHEILITIS (Gastrointestinal disorders) | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 2 | 0 | 0
DENTAL CARIES (Gastrointestinal disorders) | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 1 | 2
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 0
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 0 | 1 | 1
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 4 | 3 | 4
VOMITING (Gastrointestinal disorders) | 1 | 3 | 0
ASTHENIA (General disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 1 | 0
CHILLS (General disorders) | 0 | 0 | 1
ENERGY INCREASED (General disorders) | 0 | 1 | 0
FATIGUE (General disorders) | 9 | 6 | 6
FEELING ABNORMAL (General disorders) | 1 | 0 | 0
HUNGER (General disorders) | 0 | 0 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1 | 0
INJECTION SITE REACTION (General disorders) | 0 | 0 | 1
IRRITABILITY (General disorders) | 1 | 2 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 3 | 1 | 0
PAIN (General disorders) | 2 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 1 | 0 | 0
BODY TINEA (Infections and infestations) | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 0
FOLLICULITIS (Infections and infestations) | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1
HORDEOLUM (Infections and infestations) | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 1 | 0
TINEA PEDIS (Infections and infestations) | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 1 | 0
SUNBURN (Injury, poisoning and procedural complications) | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 0 | 0
BLOOD OESTROGEN INCREASED (Investigations) | 0 | 0 | 1
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 1 | 0 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 | 0 | 0
HEART RATE INCREASED (Investigations) | 0 | 1 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 2 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
COGNITIVE DISORDER (Nervous system disorders) | 0 | 1 | 0
COORDINATION ABNORMAL (Nervous system disorders) | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 4 | 4
DYSGEUSIA (Nervous system disorders) | 1 | 1 | 1
HEADACHE (Nervous system disorders) | 5 | 2 | 3
HYPOAESTHESIA (Nervous system disorders) | 1 | 0 | 0
LETHARGY (Nervous system disorders) | 0 | 0 | 1
MEMORY IMPAIRMENT (Nervous system disorders) | 1 | 0 | 0
MIGRAINE (Nervous system disorders) | 0 | 0 | 1
PARAESTHESIA (Nervous system disorders) | 2 | 2 | 0
POOR QUALITY SLEEP (Nervous system disorders) | 0 | 2 | 0
SINUS HEADACHE (Nervous system disorders) | 0 | 0 | 1
TREMOR (Nervous system disorders) | 1 | 0 | 0
ABNORMAL DREAMS (Psychiatric disorders) | 0 | 1 | 0
AFFECT LABILITY (Psychiatric disorders) | 1 | 0 | 0
AGITATION (Psychiatric disorders) | 1 | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 1
DEPRESSED MOOD (Psychiatric disorders) | 0 | 1 | 0
DEPRESSION (Psychiatric disorders) | 2 | 0 | 0
DISORIENTATION (Psychiatric disorders) | 0 | 1 | 0
HYPERVIGILANCE (Psychiatric disorders) | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 5 | 3 | 0
LIBIDO DECREASED (Psychiatric disorders) | 1 | 0 | 0
NERVOUSNESS (Psychiatric disorders) | 0 | 0 | 1
SLEEP DISORDER (Psychiatric disorders) | 0 | 1 | 0
DYSURIA (Renal and urinary disorders) | 2 | 1 | 0
MICTURITION URGENCY (Renal and urinary disorders) | 1 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 0
DYSPAREUNIA (Reproductive system and breast disorders) | 0 | 0 | 1
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
COLD SWEAT (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DYSHIDROSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 0 | 2
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 4 | 1 | 1
SKIN ODOUR ABNORMAL (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
FLUSHING (Vascular disorders) | 1 | 0 | 0
HOT FLUSH (Vascular disorders) | 1 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.